CLINICAL TRIAL: NCT00936520
Title: A Phase 1b, Randomized, Uncontrolled, Single-masked, Safety, Tolerability, and Pharmacokinetic Study of Multiple Doses of Three Different Concentrations (0.1%, 1.0%, 5.0%) of SAR 1118 Ophthalmic Solution in Human Subjects Undergoing Elective Pars Plana Vitrectomy (PPV)
Brief Title: SAR 1118 in Human Subjects Undergoing Pars Plana Vitrectomy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Preliminary analysis showed little or no bioactivity.
Sponsor: Johns Hopkins University (Other)
Collaborators: SARcode Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00029830
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Macular Edema (DME); Pars Plana Vitrectomy
Keywords: Diabetic Macular Edema; DME; Pars Plana Vitrectomy; Ocular Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose 1 (Experimental): SAR 1118 dose 0.1%
  Interventions: Drug: SAR 1118 0.1%
- Dose 2 (Experimental): SAR 1118 dose 1.0%
  Interventions: Drug: SAR 1118 1.0%
- Dose 3 (Experimental): SAR 1118 dose 5.0%
  Interventions: Drug: SAR 1118 5.0%

INTERVENTIONS:
Drug: SAR 1118 0.1% — Daily eye drops (twice daily, ~50 microliter [uL] each drop) approximately 10 to 12 hours apart; morning and in the evening just prior to bedtime) to the study eye only for 8 consecutive days
  Arms: Dose 1
Drug: SAR 1118 1.0% — Daily eye drops (twice daily, ~50 uL each drop) approximately 10 to 12 hours apart; morning and in the evening just prior to bedtime) to the study eye only for 8 consecutive days
  Arms: Dose 2
Drug: SAR 1118 5.0% — Daily eye drops (twice daily, ~50 uL each drop) approximately 10 to 12 hours apart; morning and in the evening just prior to bedtime) to the study eye only for 8 consecutive days
  Arms: Dose 3

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and pharmacokinetics of SAR 1118 within the anterior and posterior chamber of the eye and plasma in subjects undergoing elective vitrectomy when treated with escalating concentrations of the study drug for approximately 1 week.

DETAILED DESCRIPTION:
SAR 1118 is a potent and selective small molecule lymphocyte function antigen-1 (LFA-1) antagonist and may be therapeutically useful as a novel topical anti-inflammatory agent in a wide variety of ocular inflammatory conditions including diabetic retinopathy and diabetic macular edema. Recent evidence has demonstrated that topically delivered SAR 1118 ophthalmic solution can be detected in the aqueous, vitreous, and retina 4 to 12 hours after dosing at potentially therapeutic levels in animal models. However, the ability for the current sterile ophthalmic formulation of SAR 1118 to penetrate in sufficiently high therapeutic concentrations into the anterior and posterior chamber in humans is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Human subjects meeting the following criteria will be enrolled:

  * Age ≥18 years
  * BCVA ≤20/40 in the study eye (BCVA measured at 4M ETDRS)
  * Male or female
  * Current non-smoker (last date of smoking should be at least 60 days before study enrollment)
  * Surgically eligible to undergo elective PPV including, but not limited to, epiretinal membrane, vitreomacular traction, macular holes, or retinal detachment. The elective surgery must be able to be scheduled at least 21 days in advance to allow time for screening and for initiation of study drugs.
  * Females must be non-pregnant, non-lactating, surgically sterile for at least 3 months, post-menopausal for at least 1 years with follicle stimulating hormone (FSH) greater than or equal to 40 mIU/mL, or willing to use an approved method of contraception from 35 days prior to first study drug administration. Approved methods of contraception include: a non-hormonal intrauterine device (IUD) with spermicide, a female condom with spermicide, a diaphragm with spermicide, a cervical cap with spermicide, use of a condom with spermicide by sexual partner or sterile sexual partner.
  * Willing and able to provide written informed consent after the nature of the study has been explained, and prior to any research-related procedures.
  * Willing and able to comply with all study procedures including follow-up instructions

Exclusion Criteria:

* Individuals not eligible to participate in this study include those who meet any of the following criteria:

  * Vitreous hemorrhage
  * Active retinal detachment
  * Autoimmune disease of the anterior segment or posterior chamber including chronic keratoconjunctivitis sicca, uveitis, iritis/scleritis, blepharitis of either eye
  * Glaucoma requiring topical medications, infectious conjunctivitis, keratitis, or endophthalmitis of either eye
  * Prior vitrectomy or intraocular lens placement, within 90 days of Day 0
  * Previous intravitreal drug delivery administered in the study eye within the following time period of Day 0:

    * Intravitreal steroid given ≤3 months
    * Intravitreal vascular endothelial growth factor inhibitors given ≤2 months
  * Previous participation in any studies of investigational drugs within 1 month preceding Day 0
  * Any concurrent ophthalmic over-the-counter or topical ocular pharmaceutical within 30 days of Day 0 with the exception of saline tear lubricant.
  * History of malignancy, renal insufficiency, or hepatic insufficiency
  * Positive serum pregnancy test
  * Use of any oral, implantable, or injectable contraceptive within 30 days or 5 half-lives of the contraceptive (whichever is longer) prior to first study drug administration; patients must refrain from these types of contraceptives during the treatment period and may resume the use of such contraceptives following the 1-week observation period.
  * Any history of excessive alcohol (as judged by the Investigator) or illicit drug use/abuse
  * Consumption of any alcohol or any illicit drugs within one week of first study drug administration
  * Use of any tobacco or nicotine-containing products within 2 months prior to first study drug administration
  * Any laboratory abnormality considered clinically significant by the Investigators
  * Subjects with a hemoglobin < 12.0 g/dL
  * Any clinically significant acute or chronic medical condition that would preclude participation in a clinical study
  * Any history of autoimmune disease, immunodeficiency disorder, positive HIV, acute hepatitis A (IgM positive), or hepatitis B, or C, or organ or bone marrow transplant
  * Participation in an ongoing investigational drug or medical device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Primary outcome variable: frequency of ocular and non-ocular adverse events judged related to administration of SAR 1118 Ophthalmic Solution, or of inability to tolerate the medication. | 35 days

SECONDARY OUTCOMES:
Secondary outcome variable: concentrations of SAR 1118 in aqueous and vitreous on the day of vitrectomy. | day 9

CONTACTS AND LOCATIONS:
Overall Officials: Diana V Do, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States